CLINICAL TRIAL: NCT05536856
Title: Development and Clinical Evaluation of Topical 5-Fluorouracil Effervescent Powder Formulation in the Treatment of Vitiligo
Brief Title: Topical 5-Fluorouracil Effervescent Powder in the Treatment of Vitiligo
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35663/8/22
Record Dates: First submitted 2022-08-31; First posted 2022-09-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Vitiligo; Topical Fluorouracil; Effervescent Mixture
Keywords: Vitiligo; Fluorouracil; Effervescent powder
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): 30 patients will apply the 5-Fluorouracil plain powder on the selected patch followed by 3 milliliters of water till complete dissolution of the powder.
  Interventions: Drug: 5-Fluorouracil plain powder
- Study group (Experimental): 30 patients will apply a new effervescent mixture formula of 5-Fluorouracil prepared at faculty of pharmacy (Girls) - Al-Azhar university
  Interventions: Drug: a new effervescent mixture 5-florouracil formula

INTERVENTIONS:
Drug: a new effervescent mixture 5-florouracil formula — 30 patients will apply a new effervescent mixture 5-florouracil formula prepared at faculty of pharmacy (Girls) - Al-Azhar university
  Arms: Study group
Drug: 5-Fluorouracil plain powder — 30 patients will apply the 5-florouracil plain powder on the selected patch followed by 3 milliliters of water till complete dissolution of the powder
  Arms: Control group

SUMMARY:
A novel approach for 5-Fluorouracil delivery based on a solid effervescent formulation is proposed . 5-Fluorouracil is water soluble (~50mg/ml) and therefore has been used for the development of novel topical formulations including nano and microparticles intended for skin targeting. After hydration 5-Fluorouracil could form a complex, a suspension or even be formulated to generate effervescence. In effervescent technology, gas bubbles occur from the liquid after chemical reaction between alkali salts and organic acids (mainly citric or tartaric. Due to liberation in CO2 gas, the dissolution of drug in water is enhanced. The aim of this study is the development and clinical evaluation of topical 5-florouracil effervescent powder formulation in the treatment of vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be diagnosed as localized stable vitiligo.
* Age older than 10 years
* Stability of lesions for a duration of at least 1 year.
* Patients who didn't receive treatment for vitiligo in the previous 6 weeks before starting the study.
* Patients who agreed to join the study and signed written consent and continued till the end of the follow up period

Exclusion Criteria:

* Patients with vitiligo patches on mucous membrane,
* Patients with Koebner phenomenon,
* Other uncontrolled systemic illnesses
* Patients receiving any systemic or topical treatment for vitiligo

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Vitiligo Area Scoring Index ranged from -50 for very much worse to +50 for very much improved. Improvement means repigmentation | 3 Months
  repigmentation assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Facualty of Pharmacy, Al Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP